CLINICAL TRIAL: NCT05955625
Title: TIMELY: A Patient-centred Lifestyle Program to Support the Continuum of Care in Patients With Coronary Artery Disease Using eHealth and Artificial Intelligence
Brief Title: TIMELY: a Patient-centred Lifestyle Program for Patients With Coronary Artery Disease
Acronym: TIMELY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Collaborators: Klinik Königsfeld, Ennepetal, Germany (Unknown); Servicio Gallego de Salud (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL82723.028.23
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Coronary artery bypass graft; Lifestyle behaviour; Physical activity; Lifestyle intervention; Cardiac rehabilitation
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Because this is a behavioral intervention, the participants and clinicians cannot be blinded to the treatment condition they are randomized to. However, the evaluation of the outcome measures will be done with researchers blinded to the treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIMELY intervention and care as usual (Experimental): The intervention group will receive the TIMELY intervention including wearable monitoring devices and app in addition to care as usual for a duration of 6 months.
  Interventions: Other: TIMELY
- Care as usual (No Intervention): The care as usual group will receive the standard care as they would receive without being enrolled in the current trial.

INTERVENTIONS:
Other: TIMELY — The TIMELY app works with several devices, including a wearable activity tracker that collects activity levels, heart rate and sleep characteristics. Based on patient's activity levels, self-reported momentary mental states, health-related behaviours and environmental and clinical background factors, the app will enable patient-tailored recommendations relevant to improving lifestyle behaviours during daily life. In addition, patients will receive a blood pressure monitor that measures hemodynamic parameters through pulse wave analysis (PWA) and an easy-to-use ECG device which will be used to assess changes in heart rate and other cardiovascular measures at rest and with exercise.
  Arms: TIMELY intervention and care as usual

SUMMARY:
Study design: A randomized controlled trial will be used, where patients will be randomized (1:1) to either the control group receiving usual care or the intervention group in which patients will receive usual care in combination with the TIMELY intervention for a duration of 6 months.

Study sample: Female and male patients aged 18 years or over, with documented stable CAD and referred for cardiac rehabilitation (at > 2 weeks but <10 weeks after PCI or >4 weeks but <12 weeks after CABG or MI: STEM or non-STEMI), and/or having documented CAD by coronary angiography (stenosis in a major coronary artery >50%).

Intervention: Patients randomized to the intervention group will receive the TIMELY app on their phones or tablets for 6 months. Patients will also receive a wearable activity tracker that collects activity levels, heart rate and sleep characteristics. Based on patient's activity levels, self-reported momentary mental states, health-related behaviors and environmental and clinical background factors, the app will enable patient-tailored recommendations relevant to improving lifestyle behaviors during daily life. In addition, patients will receive a blood pressure monitor that measures hemodynamic parameters through pulse wave analysis and an easy-to-use ECG device which will be used to assess changes in heart rate and other cardiovascular measures at rest and with exercise.

Main study parameters/endpoints: The primary biomedical outcome is a change in the CoroPredict biomarker risk score from baseline (pre-randomization) to completion of the active intervention phase (6 months). The CoroPredict score is an indicator of the 10-year risk of mortality. The primary behavioral outcome is the change from baseline to 6 months in patients' functional status of fitness level (measured using the 6-minute walk test). The study further aims to improve secondary outcome measures: physical activity levels during daily life and cardiovascular responses to exercise, dietary habits, smoking behavior, medication adherence and perceived levels of psychological stress.

DETAILED DESCRIPTION:
Background of the study:

Cardiovascular diseases (CVD) are the leading cause of death globally according to the WHO. The highest burden of disease among CVDs is caused by coronary artery disease (CAD). Ageing predisposes patients to a high incidence and prevalence of CAD, in both men and women. Older patients have the greatest mortality and morbidity risk attributable to Chronic Coronary Syndromes (CCS), partially due to the high prevalence of comorbidities. Secondary prevention through comprehensive cardiac rehabilitation (CR) has been recognized as the most cost-effective intervention to limit the physiological and psychological effects of CVDs and reduce the risk of future cardiovascular events.

Contrary to pharmacological or invasive interventions for CAD, CR is far from being well implemented in all European countries and participation rates in available programs range between 30-50% of eligible patients. The TIMELY platform has been developed to stimulate a healthy lifestyle after CR. Patient-related barriers for digital health mainly involve the usability of the CR platform, especially for older patients. Thus, TIMELY includes digital tools and interfaces that will not hinder senior citizens from using them, as patient co-design has guided the development. Since lifestyle changes are key in the prevention and self-management of CAD, the main component of the TIMELY platform will be an app built on behavioral change techniques and models to empower and motivate patients to adopt a healthy lifestyle. Artificial intelligence (AI) will be employed to adapt the platform to the most current needs of the patient. In addition to prevention and self-management, the TIMELY platform will constantly monitor and predict the individual risk for disease progression or serious events and complications using validated risk scores (CoroPredict®). TIMELY will become the first AI-powered, patient-centered eHealth platform that continuously adapts and customizes CR to meet the needs of patients.

Objective of the study:

1. To investigate whether the TIMELY intervention is superior to usual care in terms of A) reducing the CoroPredict risk score (indicating risk of 10-year mortality: primary biomedical outcome) from baseline to six months; and B) increasing functional fitness levels (6-minute walk test); primary behavioral outcome) from baseline to 6 months

Study design:

A randomized controlled trial study design will be employed, where patients will be randomized (1:1) to either the control group receiving usual care or the intervention group, where patients will receive usual care in combination with the TIMELY intervention.

Assessment will take place at 4 time points: baseline, 3, 6 and 12 months post inclusion.

Patients will be asked to fill out questionnaires at 4 timepoints: baseline, 3 months, 6 months and 12 months. Through the TIMELY-platform (app) patients in the intervention group will receive prompts to conduct and ECG and blood pressure measurement. Patient in the intervention group will be wearing a Garmin, which collects information about their physical activity patterns. Lastly, patients will receive physical assessments at three time points (baseline, 6 months and 12 months), namely an exercise test and bloodwork will be done.

Study population:

Patients with documented CAD and who have been referred to cardiac rehabilitation (at > 2 weeks but < 10 weeks after PCI or > 4 weeks but <12 weeks after CABG or MI: STEMI or non-STEMI), and/or have documented CAD by coronary angiography (stenosis in a major coronary artery > 50%) will be included. Recruitment will set special focus on women, recruiting racial/ethnic minorities, older adults, rural residents, and economically disadvantaged individuals.

Intervention:

1. Timely app:

   The TIMELY app will help patients adjust their lifestyle in order for them to become healthier. The TIMELY app is supported by artificial intelligence and is based on behavioral change techniques. Through the chatbots the messages aimed at changing the behavior of patients will be personalized. Specific attention will be given to promoting physical activity. Because the chatbots can take the (physical) context of the patient into account, the odds of success are higher.
2. Wrist-worn activity tracker:

   Patients will receive an activity tracker, which will collect physical measures, such as level of activity, heart rate and sleep.
3. Tel-O-Graph:

   Patients will receive a blood pressure monitor, the Tel-O-Graph. The device additionally measures other hemodynamic parameters through pulse wave analysis (PWA).
4. Net_ECG:

   Patients will receive an easy-to-use device capable of registering atrial fibrillation.
5. eConnect HUB: Patients will receive the eConnect HUB which will transfer all data from the Tel-O-Graph to the researchers.

Patients will complete questionnaires at 4 timepoints: baseline, 3 months, 6 months and 12 months. In addition, patients will have conversations with the chatbots in the app and, based on this, receive encouragement to perform certain behaviors (e.g., exercise more or eat healthier). Through the TIMELY platform (app), patients will receive messages to take their ECG and blood pressure readings. Furthermore, patients will wear a Garmin, which will collect information about their exercise behavior. Finally, at the three measurement moments, patients will receive an exercise test. Blood will also be drawn at these times.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over (there is no a priori upper age limit)
* Documented stable CAD and referred for cardiac rehabilitation (at > 2 weeks but < 10 weeks after PCI or > 4 weeks but <12 weeks after CABG or MI: STEMI or non-STEMI) and/or having documented CAD by coronary angiography (stenosis in a major coronary artery > 50%)
* Access and ability to operate a smartphone
* Able to speak the country's native language

Exclusion Criteria:

* Unable to fully understand the provided study information and consequences of participating in the study
* Presence of a physical impairment interfering with the use of the app or devices (e.g., blindness, wheelchair bound)
* Known diagnosis of an active malignant tumour (cancer) or any other medical condition associated with a life expectancy of less than one year
* Unstable cardiovascular, cerebrovascular or other unstable medical condition
* Refusal to informed consent
* Having a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Change in risk of mortality | Baseline and 6 months
  Risk of mortality will be determined using the validated biomarker risk score CoroPredict, indicating 10-year mortality probability.
Change in functional fitness levels | Baseline and 6 months
  Functional fitness levels will be assessed using the 6-minute walking test, using the number of meters walked as the outcome.

SECONDARY OUTCOMES:
Change in physical activity | Baseline, 3 months and 6 months
  Physical activity will be measured by the validated International Physical Activity Questionnaire (IPAQ), a total score of MET minutes can be calculated.
Change in cardiovascular exercise tolerance | Baseline and 6 months
  Measures of cardiovascular responses to exercise will be based on graded symptom-limited exercise tests, using maximum watt as the outcome
Change in healthy dietary habits | Baseline, 3 months and 6 months
  Dietary habits will be assessed using the dietary questions from the validated Health Promoting Lifestyle Profiles-II questionnaire. Scores range from 9 to 36, with a higher score indicating better dietary habits.
Change in weight | Baseline and 6 months
  Weight will be measured in kilograms
Change in smoking cessation | Baseline, 3 months and 6 months
  Smoking cessation will be assessed by the validated Fagerström test. Scores range from 0-10 with a higher score indicating higher nicotine dependence.
Change in medication adherence | Baseline, 3 months and 6 months
  Medication adherence will be assessed using the validated Medication Adherence Report Scale (MARS-5) questionnaire. Scores range from 5 to 25, with a higher score indicating higher medication adherence.
Change in psychological stress levels | Baseline, 3 months, 6 months
  Psychological stress will be measured using validated the Perceived Stress Score questionnaire (PSS-10). Scores range from 0 to 40, with a higher score indicating higher levels of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jos Bosch, PhD, Principal Investigator — University of Amsterdam
Locations (3):
- Klinik Königsfeld, Ennepetal, Germany, Germany
- Willem Johan Kop, Tilburg, North Brabant, Netherlands
- Hospital Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
After trial completion, follow-up assessments, and main outcome analysis data will be (partly) available for other researchers.

REFERENCES:
- [Derived] Habibovic M, Douma E, Schafer H, Sestayo-Fernandez M, Roovers T, Sun X, Schmidt H, Kotewitsch M, Widdershoven J, Cantarero-Prieto D, Mooren F, Pena-Gil C, Gonzalez Juanatey JR, Schmidt M, Malberg H, Tsakanikas V, Fotiadis D, Gatsios D, Bosch J, Kop WJ, Schmitz B. Patient-Centered Risk Prediction, Prevention, and Intervention Platform (TIMELY) to Support the Continuum of Care in Coronary Artery Disease Using eHealth and Artificial Intelligence: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 14;14:e66283. doi: 10.2196/66283. PMID 40812736
- See also: Official website of the TIMELY project — https://www.timely-project.com/